CLINICAL TRIAL: NCT04055194
Title: Efficacy of Antenatal Tranexamic Acid in Pregnant Women With Symptomatic Placenta Previa in Decreasing Antepartum Hemorrhage - A Randomized Controlled Trial
Brief Title: Antenatal Tranexamic Acid in Women With Symptomatic Placenta Previa
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amal Ramadan, Clinical fellow of Obstetrics & Gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AntenatalTRX-PP
Record Dates: First submitted 2019-08-10; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Pregnant women with symptomatic placenta previa with previous bleeding attacks will be recruited and randomized to receive either tranexamic acid tablets (500mg four times daily) or placebo till delivery. Amount of bleeding during antepartum bleeding attacks will be estimated (by hemoglobin change from baseline at admission till delivery).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Visually-identical drug and placebo tablets will be assigned to each participant using SNOSE congaing assignment code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid group (Active Comparator): 100 pregnant women with symptomatic placenta previa with previous bleeding attacks will receive tranexamic acid tablets (500mg four times daily) till delivery.
  Interventions: Drug: Tranexamic acid tablets
- Placebo group (Placebo Comparator): 100 pregnant women with symptomatic placenta previa with previous bleeding attacks will receive placebo tablets four times daily till delivery.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Tranexamic acid tablets — Pregnant women with symptomatic placenta previa with previous bleeding attacks will receive tranexamic acid tablets (500mg four times daily) till delivery.
  Other Names: Kapron(R)
  Arms: Tranexamic acid group
Drug: Placebo oral tablet — Pregnant women with symptomatic placenta previa with previous bleeding attacks will receive placebo tablets four times daily till delivery.
  Arms: Placebo group

SUMMARY:
200 pregnant women with symptomatic placenta previa with previous bleeding attacks attending Ain Shams University maternity hospital will be recruited and randomized to receive either tranexamic acid tablets (500mg four times daily) or placebo. Amount of bleeding during antepartum bleeding attacks will be estimated (by hemoglobin change from baseline at admission till delivery).

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 28 weeks of gestation.
* Definite and reliable diagnosis of placenta previa (defined as presence of a placenta within 2 cm of the internal os), using transvaginal ultrasound scan.
* Haemodynamically stable pregnant women.
* Maternal age:20-40years old.
* Pregnant women with placenta previa, and had previous bleeding attacks or admitted with antepartum haemorrhage.

Exclusion Criteria:

* Multiple pregnancy.
* Women with bleeding tendency due to any medical disorder (ITP, thrombocytopenia, coagulopathies),or on anticoagulants .
* Severe antepartum hemorrhage and/or hemodynamic instability that necessitates urgent intervention and delivery.
* Women have hypersensitivity or any contraindication to use of tranexamic acid.
* Pregnant women with placenta previa with doppler showing morbidly adherent placenta.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Amount of bleeding during antepartum bleeding attacks | 9 weeks GA
  Amount of bleeding during antepartum bleeding attacks will be estimated by hemoglobin change from baseline at admission till delivery.

SECONDARY OUTCOMES:
Number of women requiring antepartum blood transfusion | 9 weeks GA
  Number of women requiring antepartum blood transfusion for resuscitation after severe antepartum hemorrhage.
Number of PRBCs units required during antepartum blood transfusion | 9 weeks GA
  Number of PRBCs required during antepartum blood transfusion for resuscitation after severe antepartum hemorrhage.
Number of pregnant women experiencing severe antepartum hemorrhage necessitating urgent delivery | 9 weeks GA
  Number of pregnant women experiencing severe antepartum hemorrhage necessitating urgent delivery
Gestational age at delivery | 9 weeks GA
  Gestational age in weeks at the time of delivery
Neonatal intensive care unit (NICU) admission | 9 weeks
  Number of neonates requiring NICU admission.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Ramadan, MBBCh, Principal Investigator — A Ramadan
Locations (1):
- Ain SHams Maternity Hospital, Cairo, Abbaseya, Egypt

IPD SHARING:
Plan to Share IPD: No